CLINICAL TRIAL: NCT03291093
Title: Identification of Plaque Vulnerability Wit PET/MRI: a Feasibility Study of 18F-Flutemetamol in Atherosclerosis
Brief Title: 18F-Flutemetamol and Plaque Vulnerability
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NL58543.068.16
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-01

CONDITIONS: Atherosclerosis
Keywords: PET/MRI; Amyloid; Flutemetamol
MeSH Terms: conditions — Atherosclerosis; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 18F-Flutemetamol PET/MRI dynamic (Experimental): All included patients will be patients with a recent stroke and a significant carotid plaque.
  The first 5 patients will undergo a slightly longer scan protocol to determine optimal scan time for the use of 18F-Flutemetamol in atherosclerosis imaging.
  Interventions: Drug: 18F-Flutemetamol PET/MRI
- 18F-Flutemetamol PET/MRI CEA (Experimental): 10 patients will be selected from patients that will undergo carotid endarterectomy (CEA) and will undergo the the optimized (shorter) scan protocol with 18F-Flutemetamol. The decision for this operation is made by the surgeon and neurologist and based on clinical standards and is thus independent of study participation.
  Interventions: Drug: 18F-Flutemetamol PET/MRI
- 18F-Flutemetamol PET/MRI (Experimental): The remaining 10 patients will undergo the optimized (shorter) scan protocol with 18F-Flutemetamol.
  Interventions: Drug: 18F-Flutemetamol PET/MRI

INTERVENTIONS:
Drug: 18F-Flutemetamol PET/MRI — All patients will undergo a PET/MRI of the carotids after 18F-Flutemetamol injection.

SUMMARY:
Rationale: Amyloid beta (Ab) is mainly known for its role in Alzheimer's disease (AD) pathology. However, Ab seems not only to be involved in AD pathology, but also in atherosclerosis, which might explain the remarkable similarities in risk factors between these two pathologies. In vitro studies suggest that a major part of this association is based on the ability of amyloid to lead to macrophage activation and thus inflammation. These data lead to the hypothesis that Ab is associated with plaque vulnerability.

18F-Flutemetamol is a PET tracer with high affinity for Ab. This has been extensively studied in AD patients.

Objective: To validate 18F-Flutemetamol PET in the evaluation of plaque vulnerability.

Study design: A cross-sectional validation study. Study population: 25 adults, who have recently (<14days) experienced a transient ischemic attack (TIA) or stroke with a carotid artery plaque of ≥30% and without evidence of another etiology than carotid atherosclerosis (i.e. cardiac or small vessel).

Of these 25 patients, 10 patients will be included who have been scheduled for carotid endarterectomy (CEA). The other 15 will be selected of patients who are not scheduled to undergo CEA.

Intervention: All patients will undergo a PET/MRI scan with 18F-Flutemetamol, either before the scheduled CEA or within the first 30 days following the cerebrovascular event. Imaging will include the carotid and coronary arteries as well as the brain.

Main study parameters/endpoints: Tracer uptake in the carotid artery will be correlated to vulnerable plaque characteristics as assessed by MRI. In the 10 CEA patients, tracer uptake and MR imaging of different plaque characteristics will be validated with plaque histology of the surgically removed specimen.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There is no additional benefit for study subjects. Study subjects will receive the same treatment as non-participating patients. Patients will be screened for in- and exclusion criteria to minimize risks.

For optimal MR imaging patients will be injected with a Gadolinium based contrast agent, which is a common procedure and associated with very low risk of complications. The PET tracer 18F-flutemetamol has been studied extensively and is currently used in patients with AD. Adverse events were not frequent and mainly mild. The radioactivity dose will be around 6.8 mSv.

ELIGIBILITY:
In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* All patients:

  * Age18years and older (no maximum age)
  * Informed consent by signed informed consent form regarding this study
* Patients, who are scheduled for carotid endarterectomy:

  o Inclusion criteria for carotid endarterectomy:
  * Symptomatic stenosis (TIA or CVA) within last 14days and high grade stenosis (70-99%)
  * In men, carotid artery stenosis between 50-69% is considered significant when related to clinical symptoms
* Patients, who are not scheduled for carotid endarterectomy:

  * Patients who have experienced a TIA/CVA/amaurosis fugax (a 'TIA of the eye') within the last 14 days and abnormal findings on imaging of the carotids:

    * Women with an ipsilateral carotid artery stenosis between 30-69% based on duplex ultrasonography, CTA, or MRA
    * Men with an ipsilateral carotid artery stenosis between 30-49% based on duplex ultrasonography, CTA, or MRA
    * Patients meeting inclusion criteria for carotid endarterectomy, but with contra- indications for CEA

Exclusion Criteria:

* All patients:

  * Severe cognitive impairment, neurological deficit or comorbidity causing the study to be too high a burden for the patient or disrupting patient's co- operation with scan procedures
  * Evident other causality for stroke (cardiac embolus, small vessel disease or thrombogenic diathesis)
  * Pregnant women and nursing mothers
  * Contra-indications for MRI (49):

    * Ferromagnetic implants, such as pacemakers and other electronic implants
    * Ferromagnetic (intracerebral) vascular clips
    * Metallic cochlear implants
    * Metallic splinters in eye(s) or other magnetic metallic foreign bodies elsewhere
    * Claustrophobia
  * Relative contra-indications for MRI-contrast agents (50):

    * GFR <30ml/min/1,73m2
    * Previous allergic reaction to MRI contrast agent
  * Contra-indication 18F-Flutemetamol:

    * Known allergic reaction to flutemetamol or polysorbate 80 or any of the excipients.
    * Severe liver dysfunction.
* Patients undergoing CEA:

  * Comorbidity associated with high operative risk
  * Occlusion of the internal carotid artery on the symptomatic side
  * Near occlusion on the symptomatic side
  * Complete infarction of the symptomatic anterior circulation/severe neurological deficit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
18F-Flutemetamol uptake carotids | 0-120min
  measured as SUV and TBR

SECONDARY OUTCOMES:
18F-Flutemetamol uptake coronaries | 0-150min
  measured as SUV and TBR
18F-Flutemetamol uptake in the brain | 0-150min
  measured as SUVR
CEA - plaque inflammation | 1-14 dys
  macrophage content
MRI plaque characteristics carotid | 0-150min
  semi quantitive analysis
CEA - plaque amyloid burden | 1-14 dys
  Immunohistochemistry

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Centre (MUMC+), Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided